CLINICAL TRIAL: NCT07273448
Title: Study on the Clinical Outcomes of ABO-Incompatible Living Donor Liver Transplantation
Status: Enrolling by invitation | Type: Observational
Sponsor: Ru-zhou Cai (Other)
Responsible Party: Sponsor-Investigator, Ru-zhou Cai, Principal Investigator, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Other Study IDs: BFH20251127006
Record Dates: First submitted 2025-11-20; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: ABO Incompatibility; Liver Transplant Surgery; Living Donor Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ABO-Incompatible Living Donor Liver Transplantation Patients: Evaluate the postoperative survival rate and incidence of rejection in patients undergoing ABO-incompatible living donor liver transplantation; analyze the occurrence of secondary endpoint events such as postoperative vascular complications and biliary complications; and explore relevant risk factors affecting prognosis.

SUMMARY:
Evaluate the postoperative survival rate and incidence of rejection in patients undergoing ABO-incompatible living donor liver transplantation; analyze the occurrence of secondary endpoint events such as postoperative vascular complications and biliary complications; and explore relevant risk factors affecting prognosis.

DETAILED DESCRIPTION:
Prospective and retrospective

ELIGIBILITY:
Inclusion Criteria:

1. Underwent ABO-incompatible living donor liver transplantation
2. Complete and intact clinical and follow-up data

Exclusion Criteria:

1. Non-primary liver transplantation
2. Combined other organ transplantation
3. Incomplete clinical data or loss to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients who underwent ABO-incompatible living donor liver transplantation between January 1, 2014 and December 31, 2028 and met the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative survival rate | Minimum follow-up period of 1 year postoperatively.
incidence of acute rejection | Within 1 year postoperatively

SECONDARY OUTCOMES:
Vascular complications | Within 1 year postoperatively
Biliary complications | Within 1 year postoperatively

IPD SHARING:
Plan to Share IPD: No